CLINICAL TRIAL: NCT04495673
Title: Combining Neuro-Imaging and Non-Invasive Brain Stimulation for Clinical Intervention in Opioid Use Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not reach N of participants needed
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2018-26724; 1UG3DA048508-01 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Opioid-Related Disorders; Heroin Dependence; Morphine Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence; Morphine Dependence | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tDCS with Cognitive Training (Experimental): DLPFC stimulation with tDCS with simultaneous cognitive training
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive Training
- Sham tDCS with Cognitive Training (Active Comparator): Sham tDCS with simultaneous cognitive training
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Participants receive 10 sessions (2 5-visit blocks of 46 minutes) of active tDCS to DLPFC (dorsolateral prefrontal cortex)
  Arms: tDCS with Cognitive Training
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Participants receive 10 sessions (1 5-visit block of 46 minutes of active tDCS and 1 5-visit block of sham tDCS)
  Arms: Sham tDCS with Cognitive Training
Behavioral: Cognitive Training — Executive functioning tasks

SUMMARY:
The overarching goal of this project is to expand the traditional expertise in non-invasive neuromodulation at the University of Minnesota towards developing novel paired-neuromodulation approaches using transcrancial direct current stimulation (tDCS) for new addiction treatments that support long-term abstinence. This study will investigate whether the pairing of dorsolateral prefrontal cortex (DLPFC) stimulation and cognitive training can enhance functional connectivity between DLPFC and nucleus accumbens (NAcc). We have identified higher functional connectivity between DLPFC and NAcc in alcoholics that have successfully maintained abstinence for extended periods of time (7 years). This paired-neuromodulation approach can potentially be used as a therapeutic intervention to decrease substance use probability in addiction (e.g. opioid use disorder). The long term goal is to develop new addiction treatments that support long-term abstinence in opioid use disorder. The overall objective of this proposal is to enhance functional connectivity between DLPFC and NAcc as a therapeutic intervention to enhance cognition and reduce substance use rates in opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of opioid use disorder
* Enrolled in a methadone treatment program for at least 2 months in Hennepin Healthcare and be clinically stable.
* Meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria for opioid use disorder
* Participants may have current comorbid drug use, but their primary substance use disorder diagnosis must to be based on opioid use.
* Participants must have the intention to remain in the methadone treatment program until the end of the intervention portion of the study.

Exclusion Criteria:

* Any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness>30 min, HIV)
* Head injury resulting in a skull fracture or a loss of consciousness exceeding 30 minutes (i.e., moderate or severe TBI)
* Any contraindications for tDCS or MRI scanning (tDCS contraindication: actively receiving treatment for seizures or epilepsy; MRI contraindications; metal implants, pacemakers or any other implanted electrical device, injury with metal, braces, dental implants, non-removable body piercings, pregnancy, breathing or moving disorder)
* Current active psychosis or mania
* Presence of a condition that would render study measures difficult or impossible to administer or interpret (e.g. current mania, active psychosis)
* Primary current substance use disorder diagnosis on a substance other than opioid except for caffeine or nicotine
* Current stimulant use disorder (need to be free of stimulant use for at least 1 month)
* History of electroconvulsive therapy or cortical energy exposure within the past 12 months, including participation in any other neuromodulation studies
* incarceration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lim, MD, Principal Investigator — University of Minnesota; Jazmin Camchong, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Started | 5 | 4
Completed | 3 | 2
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: (A1) Average Number of Serious Adverse Events in Active and Sham Groups.
Description: Safety was defined as the prevalence of Serious Adverse Events for the study. Subjects were monitored for Serious Adverse Events from date of first intervention session until the final follow-up visit (2 months post-intevention). Subjects were monitored using the Symptom Rating Questionnaire (SRQ), Medication/Medical Update Interview, and medical chart review. Serious Adverse Events were defined as: Death, life threatening incidents, hospitalizations (initial or prolonged), disability or permanent damage, congenital anomaly or birth defect, or an event that required intervention to prevent permanent impairment or damage. Mean and standard deviation of Serious Adverse Events was recorded across groups. A lower number indicates fewer Serious Adverse Events.
Time Frame: 2months post-intervention
Measure: Mean (Standard Deviation); unit: Number of adverse events
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 3 | 2
Number of adverse events | 0 (0) | 0 (0)

2. Primary Outcome: (A2) Activation Levels in Brain Circuits in Active and Sham Groups.
Description: Brain activation change from pre-intervention to post-intervention was planned to be compard between active tDCS and sham groups. We hypothesized that the active tDCS group will have a larger increase in brain circuit engagement than the sham group and, thus, a better outcome.
Time Frame: 1-week post-intervention
Population: Due to extreme motion artifacts preventing data acquisition, we were unable to collect minimum quantity of data necessary for the imaging analysis software to generate descriptive statistics.
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: (A3) Changes in Scaled Score on Digit Span Task.
Description: Cognitive performance change was compared between active tDCS and sham groups. Cognitive performance change was defined as improvement on the WAIS-IV Digit Span (DS). Score was calculating by subtracting the DS scaled score at baseline from the DS scaled score at 2-Month Follow Up. We hypothesized that the active tDCS group will have a larger improvement in cognitive performance than the sham group. A higher number indicates a higher impact of cognitive training and, thus, a better outcome.
  The DS Scaled Score has a range between 1 (min.) and 10 (max). Therefore, the computed difference between two DS Scaled Scores has a range of -9 (min.) to 9 (max.)
Time Frame: 2 months post-intervention
Population: Small numbers of subjects due to COVID-19 pandemic, insufficient N for interpreting data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 3 | 2
score on a scale | -2.7 (1.7) | -1.5 (1.5)

4. Primary Outcome: (A4) Number of Participants Who Relapsed After Intervention.
Description: Relapse was defined as any illiciit drug use (whether reported by the patient or reported as a positive drug screen in study or medical records) that occurred at some point between study intervention and the final follow-up visit (2 months post-intervention). Relapse was measured with the Timeline Follow Back questionnaire, saliva drug screen at the study visit, and chart review of urine drug screens. Relapse was coded 0 (did not relapse during the study) or 1 (relapsed during the study). We hypothesized that the active tDCS group will have a lower relapse rate than the sham group. A higher number indicates a higher count of participants with a relapse.
Time Frame: 2 months post-intervention
Population: Four participants who were randomized but were lost to follow-up prior to the 2 month follow up were not included in these analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 3 | 2
Participants | 2 | 0

5. Secondary Outcome: Changes in Scaled Score on Digit Symbol Task.
Description: "Durability of cognitive training was defined as improvement on the WAIS-IV Digit Scale Symbol/Coding (CD) test. The improvement period was measured between baseline and the study completion (2 months post-intervention). The score was calculated by subtracting the CD scaled score at baseline from the CD Scaled Score at 2-months post-intervention. A higher number indicates a higher impact on cognitive abilities, and a better outcome.
  The CD Scaled Score has a range between 1 (min.) and 10 (max). Therefore, the computed difference between two CD Scaled Scores has a range of -9 (min.) to 9 (max.)"
Time Frame: 2-months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
Number analyzed (Participants) | 3 | 2
score on a scale | -1 (3.6) | -1 (6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | tDCS With Cognitive Training | Sham tDCS With Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS With Cognitive Training (N=5) | Sham tDCS With Cognitive Training (N=4)
Headache (General disorders) | 1 (1) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
tingling sensation (General disorders) | 2 (3) | 1 (1)
itching sensation (General disorders) | 3 (9) | 1 (1)
burning sensation (General disorders) | 2 (7) | 0 (0)
skin redness (General disorders) | 2 (2) | 0 (0)
sleepiness/fatigue (General disorders) | 3 (6) | 1 (3)
poor concentration (General disorders) | 4 (11) | 1 (2)
acute mood change (General disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT04495673/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04495673/ICF_001.pdf